CLINICAL TRIAL: NCT03602625
Title: Risk Factors of Preterm Birth Born in Hospital：a Prospective Multicenter Case-control Study
Acronym: RFPTB
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: EKYYRFPTBMC
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Risk Factors
Keywords: Premature birth; Risk factors
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm group: All the live-born infants with gestational age less than 37weeks and more than 20weeks born in the cooperative hospital every day or every two or three days.
- Term group: The one next-live-born infants with gestational age at 37weeks or more than 37weeks.

SUMMARY:
The purpose of this study is to explore the perinatal risk factors of preterm birth in China.

DETAILED DESCRIPTION:
Preterm birth is a global scourge, and the leading cause of newborn deaths (babies in the first 4 weeks of life) and raised to the leading cause of death among children under 5 years of age, responsible for approximately 1 million deaths in 2015. In China, the prevalence of preterm increased from 4~5% in 1990s to 7~10% in 2010. Preterm birth become a burden to both the family and society. Therefore, the risk factors of preterm birth become the critical issue of both Obstetrics and Neonatology. More importantly, few multicenter prospective studies on risk factors of preterm birth included potential reasons such as maternal occupation, psychology condition and lifestyles during pregnancy were conducted in China. Thus, the aim of our study is to explore the perinatal risk factors of preterm birth nowadays in China.

ELIGIBILITY:
Inclusion Criteria:

* Live-born infants >20weeks of gestational age

Exclusion Criteria:

* Stillbirth

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Live-born preterm infants and one term infants born following the preterm infants in the same cooperation hospitals
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
live-born preterm | at birth
  less than 37weeks gestational age

SECONDARY OUTCOMES:
birth weight (g) | at birth
  Infant's weight recorded at the time of birth
gestation age (week) | at birth
  the number of completed weeks of gestation, which was determined by the duration of menorrhoea or confirmed by an early ultrasound scan during pregnancy
Apgar score | 1min after birth
  determined by evaluating the newborn baby on five simple criteria（Appearance, Pulse, Grimace, Activity, Respiration） on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10.
Apgar score | 5min after birth
  determined by evaluating the newborn baby on five simple criteria（Appearance, Pulse, Grimace, Activity, Respiration） on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10.
small for gestational age | at birth
  a birth weight below the 10th percentile for the gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chao, PhD, MD, Study Director — Children's Hospital of Fudan University
Locations (15):
- China (15):
  - Xiamen Maternal and Child Health Care Hospital, Xiamen, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Maternal and Child Health Hospital of Hainan Province, Haikou, Hainan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Changzhou Maternal and Child Health Care Hospital, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Tongxin County People's Hospital, Wuzhong, Ningxia
  - The First People's Hospital of Yinchuan, Yingchuan, Ningxia
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Jining NO.1 People's Hospital, Jining, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Jimo People's Hospital, Qingdao, Shandong
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Songjiang Maternity & Child Health Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Yueqing Hospital Affiliated to Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu L, Oza S, Hogan D, Chu Y, Perin J, Zhu J, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of under-5 mortality in 2000-15: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet. 2016 Dec 17;388(10063):3027-3035. doi: 10.1016/S0140-6736(16)31593-8. Epub 2016 Nov 11. PMID 27839855
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- See also: A prospective multicenter epidemiology investigation of premature newborn — http://kns.cnki.net/KCMS/detail/detail.aspx?FileName=1013103173.nh&DbName=CDFD2013
- See also: Prevalence of singleton preterm birth in 10 cities of China in 1993-2005 — http://kns.cnki.net/KCMS/detail/detail.aspx?FileName=ZHLX200711005&DbName=CJFQ2007